CLINICAL TRIAL: NCT04270383
Title: A Multicenter Observational Study About the Clinical Characteristics and Long-term Prognosis of 2019-nCoV Infection in Children
Brief Title: Clinical Characteristics and Long-term Prognosis of 2019-nCoV Infection in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Capital Institute of Pediatrics, China (Other); The First Affiliated Hospital of Anhui Medical University (Other); China-Japan Friendship Hospital (Other); The First Affiliated Hospital of Xiamen University (Other); Guangzhou Women and Children's Medical Center (Other); Shenzhen Children's Hospital (Other Government); First Affiliated Hospital of Guangxi Medical University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Hainan People's Hospital (Other); Children's Hospital of Hebei Province (Other); Wuhan Women and Children's Medical Center (Other); Changchun Children's Hospital (Other); Children's Hospital of Nanjing Medical University (Other); Jiangxi Province Children's Hospital (Other); Shengjing Hospital (Other); Shanxi Provincial Maternity and Children's Hospital (Other); Xian Children's Hospital (Other Government); Children's Hospital of Chongqing Medical University (Other); Tianjin Children's Hospital (Other); Tianjin Medical University Second Hospital (Other); Kunming Children's Hospital (Other); Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Kunling Shen, Director of National Clinical Research Center for Respiratory Diseases, China, Beijing Children's Hospital
Other Study IDs: BCH Lung 012
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: 2019-nCoV
Keywords: 2019-nCoV infection; 2019-nCoV pneumonia; Children
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2019-nCoV infection group: Children hospitalized with direct laboratory confirmed of novel coronavirus with or without pneumonia are classified as the 2019-nCoV infection group.
- Control group: Children hospitalized with pneumonia other than the novel coronavirus pneumonia during the same hospitalization period as 2019-nCoV infection group are classified as the control group.

SUMMARY:
The study is designed to clarify the clinical characteristics, risk factors and long-term prognosis of children with 2019-nCoV infection in China.

DETAILED DESCRIPTION:
As of February 10th, 2020, more than 40,000 human have been confirmed infected with a novel coronavirus (2019-nCoV) in China, with at least 800 reported deaths. Additional cases have been confirmed in multiple countries, and some are reported in children. Patients with confirmed 2019-nCoV infection have reported respiratory illness with fever, cough, et al. Some are asymptomatic carriers. However, there are relatively few diagnosed cases of children, and the long-term prognosis is unknown. Therefore, a multicenter observational study is needed to better understand the clinical characteristics of 2019-nCoV infection in children.

This observational study will last from February to December 2020. The patients enrolled were diagnosed with 2019-nCoV infection or 2019-nCoV pneumonia by Beijing Children's Hospital and other members of Chinese National Clinical Research Center for Respiratory Diseases in 2019-2020. At the same time, children hospitalized with pneumonia other than 2019-nCoV pneumonia during the same period are classified as the control group by 3~5:1 matching for age and sex to the 2019-nCoV group. After guardians signing the informed consent forms, all the participants' clinical data, laboratory examination results, image data and also the follow-up information after six months of their treatment will be collected.

The trial will be completed in 10 months, with subjects recruited from the hospitals that in partnership with clinical research collaboration of National Clinical Research Center for Respiratory Diseases.

ELIGIBILITY:
1. For the 2019-nCoV infection group

   Inclusion Criteria:

   Diagnosed with 2019-nCoV infection (with direct laboratory evidence).
   1. Respiratory or blood samples tested positive for novel coronavirus nucleic acid with RT-PCR.
   2. Gene sequencing of respiratory or blood samples show highly homologous with known novel coronaviruses.

   Exclusion Criteria:

   Subjects will be excluded if the children or their parents disagree to conduct this study.
2. For the control group

Inclusion Criteria:

1. Diagnosed with pneumonia, and excepted of novel coronavirus infection.
2. The hospitalization time is the same as that of novel coronavirus pneumonia.

Exclusion Criteria:

Subject will be excluded if she or he has one of the following:

1. First diagnosis is not pneumonia.
2. Any one of the novel coronavirus laboratory test results show positive.
3. Children or their parents disagree to conduct this study.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who are aged 1day to 18 years, and diagnosed with 2019-nCoV infection/pneumonia or pneumonia other than novel coronavirus hospitalized in the same period in China.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-02-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The cure rate of 2019-nCoV. | 6 months
  Percentage
The improvement rate of 2019-nCoV. | 6 months
  Percentage
The incidence of long-term adverse outcomes. | 6 months

SECONDARY OUTCOMES:
Duration of fever | 2 weeks
  Days
Duration of respiratory symptoms | 2 weeks
  Days
Duration of hospitalization | 2 weeks
  Days
Number of participant(s) need intensive care | 2 weeks
Number of participant(s) with acute respiratory distress syndrome | 2 weeks
Number of participant(s) with extra-pulmonary complications, including shock, renal failure, multiple organ failure, hemophagocytosis syndrome, et al. | 2 weeks
Number of participant(s) who died during the trial | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Kunling Shen, MD,PhD, Principal Investigator — Beijing Children's Hospital of Capital Medical University, China; Tianyou Wang, MD,PhD, Principal Investigator — Beijing Children's Hospital of Capital Medical University, China; Baoping Xu, MD,PhD, Principal Investigator — Beijing Children's Hospital of Capital Medical University, China
Locations (1):
- Beijing Children's Hospital,, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided